CLINICAL TRIAL: NCT01766128
Title: Randomized Double Blind Placebo-controlled Study of Zonisamide Effectiveness in Early Parkinson Disease
Brief Title: Study of Zonisamide in Early Parkinson Disease
Acronym: ZONIST
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Practical problems
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasim Tabrizi, Assistant professor of neurology, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZEPD-1091
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Early stage; Zonisamide; UPDRS
MeSH Terms: conditions — Parkinson Disease | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zonisamide (Active Comparator): The patients in this arm are treated with zonisamide 50mg/d
  Interventions: Drug: Zonisamide
- Placebo (Placebo Comparator): The patients in this arm are treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide — The first arm will be treated by zonisamide
  Arms: Zonisamide
Drug: Placebo — The second arm will receive placebo
  Arms: Placebo

SUMMARY:
The aim of this study is investigation of neuroprotective effect of zonisamide in early Parkinson disease. A total of 60 patients with early Parkinson disease who meet the study criteria will be enrolled and randomized into two groups alternately based on their visit date. Demographic data, Unified Parkinson's Disease Rating Scale (UPDRS), modified Hoehn&Yahr and modified Schwab&England activities of daily living scale will be determined and registered for each patient. Patients of group A will be treated by zonisamide 50mg/d for 12 months and the other group will be treated by placebo for the same time. Primary endpoint is occurrence of parkinsonian symptoms which interfere with patients' daily activity or cause psychosocial embarrassment. The mentioned scores will be registered every 2 months for both groups by blinded neurologist and also regular blood test will be performed to prevent drug adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-85 years
2. Symptoms and signs of idiopathic Parkinson disease for less than a month that do not lead to physical or psychosocial disability.

Exclusion Criteria:

1. Past history of treatment with antiparkinson drugs.
2. Past history of treatment with zonisamide
3. Hepatic insufficiency (ALT>2ULN)
4. Renal insufficiency (Cr>2mg/dl)
5. Self or family history of nephrolithiasis
6. Active psychosis
7. Epilepsy
8. Suicidal attempt in last 3 years
9. Hypersensitivity to sulfonamides
10. Pregnancy and breastfeeding

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Time to need for dopaminergic therapy | Baseline and month 6

SECONDARY OUTCOMES:
change in UPDRS score | Baseline and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Etemadifar, Principal Investigator — IUMS